CLINICAL TRIAL: NCT00941616
Title: An Open-label, Multi-centre Study to Assess the Pharmacokinetics, Efficacy and Safety of Biostate® in Subjects With Von Willebrand Disease.
Brief Title: Study of a pd VWF/FVIII Concentrate, Biostate®, in Subjects With Von Willebrand Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-08-54; 1481 (Other: CSL Behring); 2008-004922-18 (EudraCT Number)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Von Willebrand Disease
Keywords: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; von Willebrand Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PK (Experimental): Includes subjects participating in the pharmacokinetic component of the study.
  Interventions: Biological: Biostate®
- Prophylaxis (Experimental): Includes subjects receiving 12 months of prophylactic therapy.
  Interventions: Biological: Biostate®
- On-demand (Experimental): Includes subjects receiving 12 months of on-demand treatment.
  Interventions: Biological: Biostate®
- Cross-over to prophylaxis (Experimental): Includes subjects completing 12 months of on-demand treatment (the "On-demand" arm) who cross-over to prophylactic therapy for an additional 12-month period.
  Interventions: Biological: Biostate®

INTERVENTIONS:
Biological: Biostate® — 80 IU vWF/kg administered as a bolus intravenous infusion on Day 1 and approximately Day 180
  Other Names: Human Coagulation Factor VIII / von Willebrand Factor
  Arms: PK
Biological: Biostate® — Frequency and dose will be determined by the Investigator based on the subjects clinical condition, previous VWF concentrate requirements, response to therapy, weight and reason for usage.
  Other Names: Human Coagulation Factor VIII / von Willebrand Factor
  Arms: Cross-over to prophylaxis; On-demand; Prophylaxis

SUMMARY:
The aim of this study is to assess the pharmacokinetics (PK), efficacy, and safety of Biostate® in subjects with Von Willebrand Disease (VWD).

Pharmacokinetic Component:

PK parameters will be determined from a subgroup of subjects. Subjects who complete the PK component will subsequently continue in the efficacy component of the study, either continuing on a previously established prophylaxis regimen or continuing to receive on-demand treatment with the occurrence of non-surgical bleeding (NSB) events.

Efficacy Component:

Three treatment arms are defined for the efficacy component of the study. (1) Subjects who are currently being treated on a set prophylaxis regimen with a VWF product at the time of study entry will be enrolled in the "Prophylaxis" arm. (2) Subjects not being treated on a set prophylaxis regimen at the time of study entry who require a VWF product for the treatment of NSB events will be enrolled in the "On-demand" arm and commence using Biostate in the treatment of NSB events. (3) Subjects enrolled in the "On-demand" arm have the possibility to enter the "Cross-over to Prophylaxis" arm to receive an additional 12 months of prophylactic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with VWD
* Desmopressin acetate (DDAVP) treatment is ineffective or contraindicated or not available
* Evidence of vaccination against hepatitis A and B (or presence of antibodies against hepatitis A and B) within 10 years prior to their first dose of Biostate®
* Written informed consent given

Exclusion Criteria (for participation in the PK component):

* Actively bleeding immediately prior to initial PK period
* Have received DDAVP or a VWF product in the 5 days prior to their first dose of study product
* Have Type 2B, 2N or 2M VWD

Exclusion Criteria (for all subjects):

* Requiring a VWF product for a planned surgical procedure at enrolment
* Have received aspirin or other non-steroidal anti-inflammatory drugs within 7 days prior to their first dose of study product
* Known history of, or are suspected to have, VWF or FVIII inhibitors
* Suffering an acute or chronic medical condition, other than VWD, which may affect the conduct of the study
* Known or suspected hypersensitivity or previous evidence of severe side effects to Biostate®, VWF/FVIII concentrates, or human albumin
* Impaired liver function at screening
* Evidence or a history (within the previous 12 months) of abuse of any drug substance, licit or illicit
* Participation in a clinical study or use of an investigational compound in the 3 months preceding the first day of study drug administration, or plans to enter such a study during the study period.
* Females who are pregnant, breast-feeding or who have a positive pregnancy test at screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Haemostatic efficacy at time of non-surgical bleeding (NSB) event | From Day 1 until final study visit
Haemostatic efficacy overall | Monthly (prophylactic therapy) or once every 3 months (for on-demand use)
Number of treatments with blood product transfusions required to resolve any bleeding event | From Day 1 until final study visit
vWF/FVIII concentrate usage (number of infusions, IU/kg per dose, per event, per month and per year) | From Day 1 until final study visit
Assessment of blood loss during any surgical procedure | From Day 1 until final study visit
Number of spontaneous or traumatic NSB events | From Day 1 until final study visit
Pharmacokinetic parameters for vWF and FVIII (PK arm only) | Up to 72 hours following infusions on Day 1 and approximately Day 180

SECONDARY OUTCOMES:
Development of FVIII inhibitors | From Day 1 until final study visit
Development of vWF inhibitors | From Day 1 until final study visit

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (5):
- Study Site, Sofia, Bulgaria
- Poland (2):
  - Study Site, Warsaw
  - Study Site, Wroclaw
- Study Site, Barnaul, Russia
- Study Site, Lviv, Ukraine